CLINICAL TRIAL: NCT03700749
Title: Pragmatic Multicentre FActorial Randomised Controlled triaL Testing Measures to reduCe Surgical Site Infection in lOw and Middle Income couNtries
Brief Title: FALCON Trial Testing Measures to Reduce Surgical Site Infection
Acronym: FALCON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Lagos State University (Other); Universidad Francisco Marroquín (Other); Kigali University Teaching Hospital (Other); Christian Medical College and Hospital, Ludhiana, India (Other); University of Edinburgh (Other); University of the Philippines (Other); King Edward Medical University (Other); University of Witwatersrand, South Africa (Other); Universidad Peruana Cayetano Heredia (Other); Centre National Hospitalier Universitaire (Unknown); Ndola Teaching Hospital (Unknown); Hospital Espanol de Veracruz (Unknown); Ministry of Health, Ghana (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RG_17-126
Record Dates: First submitted 2018-08-23; First posted 2018-10-09 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Abdominal Surgery; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: FALCON 2x2 factorial trial with strata: (1) clean-contaminated and (2) contaminated/dirty. Eligible patients will be randomised at the level of the individual in a 1:1:1:1 ratio between:
  A. 2% alcoholic chlorhexidine and non-coated suture B. 2% alcoholic chlorhexidine and triclosan-coated suture C. 10% aqueous povidone-iodine and non-coated suture D. 10% aqueous povidone-iodine and triclosan-coated suture
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded. The operating surgeon will not perform outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2%chlorhexidine + non-coated suture (Active Comparator): 2%alcoholic chlorhexidine + non-coated suture. Intervention: skin preparation with 2%alcoholic chlorhexidine in combination with non-coated suture for abdominal fascial closure.
  Interventions: Drug: 2% chlorhexidine + non-coated suture
- 2%chlorhexidine + coated suture (Active Comparator): 2%alcoholic chlorhexidine + triclosan-coated suture. Intervention: skin preparation with 2%alcoholic chlorhexidine in combination with triclosan-coated suture for abdominal fascia closure.
  Interventions: Drug: 2% chlorhexidine + coated suture
- 10% povidone-iodine + non-coated suture (Active Comparator): 10% povidone-iodine and non-coated suture. Intervention: skin preparation with 10% povidone-iodine in combination with non-coated suture for abdominal fascial closure.
  Interventions: Drug: 10%povidone-iodine + non-coated suture
- 10%povidone-iodine + coated suture (Active Comparator): 10%povidone-iodine/triclosan-coated suture. Intervention: skin preparation with 10% povidone-iodine in combination with triclosan-coated suture for abdominal fascial closure.
  Interventions: Drug: 10%povidone-iodine + coated suture

INTERVENTIONS:
Drug: 2% chlorhexidine + non-coated suture — Interventions:
  2% alcoholic chlorhexidine non-coated suture
  Arms: 2%chlorhexidine + non-coated suture
Drug: 2% chlorhexidine + coated suture — Interventions:
  2% alcoholic chlorhexidine triclosan coated suture
  Arms: 2%chlorhexidine + coated suture
Drug: 10%povidone-iodine + non-coated suture — Interventions:
  10% povidone-iodine non-coated suture non-coated suture
  Arms: 10% povidone-iodine + non-coated suture
Drug: 10%povidone-iodine + coated suture — Interventions:
  10% povidone-iodine triclosan coated suture
  Arms: 10%povidone-iodine + coated suture

SUMMARY:
FALCON is a Pragmatic multi-centre trial testing measures to reduce superficial or deep skin infection following abdominal surgery in low and middle income countries. The trial will recruit patients undergoing abdominal surgery. Recruited participants will be randomly assigned to four arms to receive different combinations of skin preparation and sutures for would closure:

A. In this arm surgeon will use 2% alcoholic chlorhexidine for skin cleansing and non-coated suture for wound closure; B. In this arm surgeon will use 2% alcoholic chlorhexidine for skin cleansing and triclosan coated suture for wound closure; C. In this arm surgeon will use for operation 10% aqueous povidone-iodine for skin cleansing and non-coated suture for wound closure; D. In this arm surgeon will use 10% aqueous povidone-iodine for skin cleansing and triclosan-coated suture.

DETAILED DESCRIPTION:
FALCON is a pragmatic, blinded (patient and outcome assessor), 2x2 factorial, stratified, multi-centre randomised controlled trial, with an internal pilot, to evaluate measures to reduce Surgical Site Infection (SSI) rates in patients undergoing surgery with an abdominal incision.

Surgical site infection (SSI) represents a major burden for patients, doctors, and health systems across all settings. SSI is the commonest postoperative complication worldwide and the commonest healthcare-associated infection in low and middle income countries (LMICs). SSIs cause pain, discomfort, disability, and increase the time taken to return to work (3). SSIs increase healthcare costs in all health settings. Whilst there is no direct data on the costs of SSI in LMICs, within the UK National Health Service, SSIs cost approximately £3500 per patient and £700 million per year in total. The impact of increased healthcare costs on patients, communities, and providers can be major in LMICs where personal income is low and patients may be required to pay for their own treatment. SSI has also been associated with one-third of postoperative deaths and accounts for 8% of all deaths caused by a hospital acquired infection.

Strata in FALCON trial are defined according to the anticipated category of wound contamination: (1) clean-contaminated and (2) contaminated/dirty. Eligible patients will be randomised at the level of the individual in a 1:1:1:1 ratio between:

A. 2% alcoholic chlorhexidine and non-coated suture B. 2% alcoholic chlorhexidine and triclosan-coated suture C. 10% aqueous povidone-iodine and non-coated suture D. 10% aqueous povidone-iodine and triclosan-coated suture.

Participant will be recruited from hospitals in Low and Middle Income Countries (LMICs). Participants who is undergoing abdominal surgery with an anticipated clean-contaminated, contaminated or dirty surgical wound will be selected to enter the trial.

The 6 month internal pilot will assess the feasibility of recruitment, compliance with treatment allocation and patient retention and follow-up rates. The main RCT will recruit 5480 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one abdominal incision that is ≥5cm (open or laparoscopic extraction site), with an anticipated clean-contaminated, contaminated or dirty surgical wound.
* Patients undergoing emergency (surgery on an unplanned admission) or elective (surgery on a planned admission) operations.
* Any operative indication, including trauma surgery.
* Patient able and willing to provide written informed consent (signature or a fingerprint).
* Paediatric and adult patients. This criteria is made country-specific. Each country decides the lower age limit for the trial. This is dependent on country-specific regulatory approvals. Age eligibility will vary by country.

Exclusion Criteria:

* Patients with a documented or suspected allergy to iodine, shellfish, or chlorhexidine skin preparation solution.
* Patient unable to complete post-operative follow-up (i.e. will not be contactable after discharge).

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5480 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection (SSI) | At 30-days post-surgery
  Deep incisional or superficial incisional SSI which must occur within 30 days of the index operation. The infection must involve the skin, subcutaneous, muscular or fascial layers of the incision. Patient must at least have one of the following: (1) purulent discharge from wound; (2) organisms detected from wound swab; (3) Wound opened spontaneously or by a clinician AND, at the surgical wound, the patient has at least one of: pain or tenderness; localised swelling; redness; heat; systemic fever (>38°C); (4) Diagnosis of SSI by a clinician or on imaging.

SECONDARY OUTCOMES:
Physiological parameter - SSI at discharge from hospital | Within 30-days post surgery from index operation
  Deep incisional or superficial incisional SSI. The infection must involve the skin, subcutaneous, muscular or fascial layers of the incision and the patient must have one of the following: (1) purulent discharge from wound; (2) organisms detected from wound swab; (3) Wound opened spontaneously or by a clinician AND, at the surgical wound, the patient has at least one of: pain or tenderness; localised swelling; redness; heat; systemic fever (>38°C); (4) Diagnosis of SSI by a clinician or on imaging.
Mortality - patient mortality status | Within 30-days post surgery from index operation
  Mortality within 30-days post surgery
Physiological parameter - Unplanned wound opening | Within 30-days post surgery from index operation
  Whether an unplanned wound opening has occurred at abdominal surgical site within 30-days post surgery, spontaneously opened or by clinician
Re-operation for SSI | Within 30-days post surgery from index operation
  Re-operation for SSI within 30-days post surgery
Length of hospital stay for index admission | Within 30-days post surgery from index operation
  Length of hospital stay for index admission will be collected and will measure time from surgery to time of discharge.
Participant's Readmission | Within 30-days post surgery from index operation
  Whether patient readmitted within 30-days post surgery
Questionnaire - return to normal activities | Within 30-days post surgery from index operation
  Return to normal activities (e.g. work, school, or family duties) ascertained by trial specific questionnaire
Resistance of organisms | Within 30-days post surgery from index operation
  Resistance of organisms detected from wound swabs to prophylactic antibiotics administered within 1 hour of incision
Questionnaire - Health resource usage | Within 30-days post surgery. Health resource usage will only be collected for adult patients (aged 18 and above) at pre-selected centres. This will include costs of post-operative visits to various healthcare professionals.
  Health resource usage within 30-days post surgery ascertained by trial specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dion Morton, Principal Investigator — University of Birmingham
Locations (1):
- Lagos University Teaching Hospital, Lagos, Nigeria

REFERENCES:
- [Derived] NIHR Global Health Research Unit on Global Surgery. Mechanisms and causes of death after abdominal surgery in low-income and middle-income countries: a secondary analysis of the FALCON trial. Lancet Glob Health. 2024 Nov;12(11):e1807-e1815. doi: 10.1016/S2214-109X(24)00318-8. Epub 2024 Sep 5. PMID 39245053
- [Derived] NIHR Global Health Research Unit on Global Surgery. Accuracy of the Wound Healing Questionnaire in the diagnosis of surgical-site infection after abdominal surgery in low- and middle-income countries. Br J Surg. 2024 Jan 31;111(2):znad446. doi: 10.1093/bjs/znad446. PMID 38747515
- [Derived] Monahan M, Glasbey J, Roberts TE, Jowett S, Pinkney T, Bhangu A, Morton DG, de la Medina AR, Ghosh D, Ademuyiwa AO, Ntirenganya F, Tabiri S; NIHR Global Research Health Unit on Global Surgery. The costs of surgical site infection after abdominal surgery in middle-income countries: Key resource use In Wound Infection (KIWI) study. J Hosp Infect. 2023 Jun;136:38-44. doi: 10.1016/j.jhin.2023.03.023. Epub 2023 Apr 21. PMID 37086854
- [Derived] NIHR Global Research Health Unit on Global Surgery. Routine sterile glove and instrument change at the time of abdominal wound closure to prevent surgical site infection (ChEETAh): a pragmatic, cluster-randomised trial in seven low-income and middle-income countries. Lancet. 2022 Nov 19;400(10365):1767-1776. doi: 10.1016/S0140-6736(22)01884-0. Epub 2022 Oct 31. PMID 36328045
- [Derived] NIHR Global Research Health Unit on Global Surgery. Reducing surgical site infections in low-income and middle-income countries (FALCON): a pragmatic, multicentre, stratified, randomised controlled trial. Lancet. 2021 Nov 6;398(10312):1687-1699. doi: 10.1016/S0140-6736(21)01548-8. Epub 2021 Oct 25. PMID 34710362